CLINICAL TRIAL: NCT03803839
Title: Could the Intra-operative Clodronate Rinsing Improve the Integration of the Femoral Stem in a Prospective, Double-blinded, Randomized, Placebo-controlled Clinical RSA-study
Brief Title: Locally Administered Clodronate in the Prevention of Aseptic Implant Loosening
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Oulu (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Ei tiedossa
Record Dates: First submitted 2019-01-04; First posted 2019-01-15 (Actual); Last update posted 2019-01-18 (Actual); Status verified 2019-01

CONDITIONS: Hip Arthrosis
Keywords: RSA; DXA; Bisphosphonates; Migration of stem; Aseptic loosening of prosthesis
MeSH Terms: conditions — Osteoarthritis, Hip | interventions — Clodronic Acid; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: In this prospective, double-blinded, randomized, placebo-controlled clinical trial with two years follow-up period the investigators rinsed the proximal intramedullary cavity of the femur with either clodronate (60 mg clodronate in 1000 ml saline) or saline (1000 ml saline) prior to the application of the femoral stem.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Patients were randomized into two treatment groups; either the clodronate or a placebo group. All patients, surgeons and other personnel in the operating theatre were blinded as to the patients' study group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Clodronate (Active Comparator): 1 mM clodronate (60 mg in 1000 ml saline) was used intraoperatively during total hip arthroplasty: before installation of the prosthesis, the rinsing was performed with pulsatile lavage using the clodronate solution. The time for rinsing was about one minute.
  Interventions: Drug: Clodronate
- Saline (Placebo Comparator): 1000 ml saline was used intraoperatively during total hip arthroplasty: before installation of the prosthesis, the rinsing was performed with pulsatile lavage using the saline solution. The time for rinsing was about one minute.
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Clodronate
  Arms: Clodronate
Drug: Saline
  Arms: Saline

SUMMARY:
Periprosthetic bone-loss after total hip arthroplasty (THA), detected as an early migration of the prosthesis, may predict later loosening. The investigators hypothesized that by reducing bone resorption after THA with bisphosphonates, it might be possible to achieve better early fixation of the implant.

Nineteen patients suffering arthrosis were recruited to a prospective, double-blinded, randomized, placebo-controlled clinical pilot trial. Patients were operated with an uncemented Bimetric stem with tantalum markers, the acetabular cup and liner were chosen by the surgeon. The femoral proximal intramedullary canal was rinsed with 1mM (millimole) clodronate, that was done by adding the clodronate to the 1000 ml 0.9% NaCl (sodium chloride) in nine patients and rinsing solution was the pure 0.9% NaCl for 10 patients. These rinsing packages were labeled only with the code from the pharmacy of the hospital. These patients were followed for two years using radiostereometric analysis (RSA), dual energy x-ray absorptiometry (DXA) and the Harris hip score (HHS).

The purpose of the investigator's study was to examine whether the local intraoperative administration of clodronate could reduce periprosthetic bone loss and further stem migration after primary THA.

ELIGIBILITY:
Inclusion Criteria:

* hip arthrosis and
* a primary THA was planned

Exclusion Criteria:

* renal insufficiency
* hypercalcemia
* malignant tumors
* contemporaneously treatment with another bisphosphonate or aminoglycoside

Max Age: 73 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2004-03-26 (Actual); Primary Completion 2014-03-12 (Actual); Study Completion 2014-03-12 (Actual)

PRIMARY OUTCOMES:
Maximal total point motion (MTPM) - migration of the femoral stem | 0 to 24 months
  It represents the length of the translation vector of the point in a rigid body that has the greatest motion. It can only have positive values, and is not normally distributed. The reason for using MTPM is that in many cases, motion implies a biological effect of some kind and this effect is liable to be greatest at the point of maximum motion. The parameter has been measured by RSA-methods, which is an accurate method of determining the migration and wear of orthopaedic implants: it determine the precise location of two distinct objects relative to each other in three dimension such as the relative position of the femoral component and the proximal femur. In radiostereometric analysis the position in space of the original object is reconstructed from a two dimensional x-ray film using tantalum beads. Movement between segments is then calculated by localizing each segment in a coordinate system. Lower values represent a better outcome.

SECONDARY OUTCOMES:
Bone mineral density (BMD) in 7 Gruen zones | 0 to 24 months
  BMD was measured by dual-energy X-ray absorptiometry, DXA. In clinical use, precision errors are < 5 %. To evaluate the horizontal linear distribution of the BMD, seven Gruen zones, peri-prosthetic sub-regions of interest, ROI (region of interest) were calculated by the software on the anteroposterior view of the proximal femur. The value of BMD is g/cm2 and it estimates the strength of the bone. Higher values/lesser decrease in values represent a better outcome.

OTHER OUTCOMES:
Migration of femoral stem | 0 to 24 months
  Subsidence and vertical movement of the femoral stem (scale micrometers), x-, y- and z-translations. Parameters were measured using RSA-methods and the scaling is linear. Lower values represent a better outcome.
The maximal (MTPM) maximal total point motion | 3 to 24 months
  The maximal MTPM value after 3 months when the expected integration of stem should have happened. Lower values represent a better outcome.
Correlation between baseline BMD and the maximal MTPM | BMD (0 month) - the maximal MTPM 3 to 24 months
  This parameters summarize the BMD and RSA values together. The investigators have planned it to evaluate the correlation between the quality of periprosthetic bone in baseline and the migration of femoral stem during 2 years follow-up period between the study groups.
Harris Hip Score (HHS) | 0 to 24 months
  Harris Hip Score (HHS) is a clinician-based outcome measure, health status scale, that is frequently used to measure the outcome of total hip arthroplasty. It is measured by questionnaire that give points from 0 to 100. Higher values represent a better outcome.

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary and secondary outcome data will be made available.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available after submitting the results to the scientific journals and five years after the publication.
Access Criteria: Data Access requests will be reviewed By an external Independent Review Panel. Requestors will be required to sign a Data Access Agreement.